CLINICAL TRIAL: NCT06927050
Title: Visual Communication: Can a Digital Tool Improve the Understanding of Treatment Options for Patients With Cancer and Increase Satisfaction of the Overall Experience for Patients, Caregivers, and Providers?
Brief Title: Visual Communication: Digital Tool to Improve the Understanding of Treatment Options for Patients With Cancer and Increase Satisfaction of the Overall Experience for Patients, Caregivers, and Providers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-01870
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (and caregivers) recently diagnosed with cancer (Experimental): Enrolled patients will receive a tool during the patient consultation encounter to explain their disease location and stage, role of radiation, logistics of radiation treatment delivery and sequencing of treatment. Following the encounter, a survey will be provided.
  If patients are accompanied by a caregiver(s), they will also receive a survey.
  Interventions: Behavioral: Visual Communication Tool

INTERVENTIONS:
Behavioral: Visual Communication Tool — MyCareGorithm will be used during the patient consultation encounter to explain their disease location and stage, role of radiation, logistics of radiation treatment delivery and sequencing of treatment. MyCareGorithm is an online educational tool that will be displayed to the patient via iPad or Microsoft tablet.
  Other Names: MyCareGorithm

SUMMARY:
This is a study in patients with newly diagnosed cancer to prospectively evaluate the feasibility of integration of a visual communication tool for patients/caregivers/providers by determining whether such a tool can increase overall satisfaction with the patient experience.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Patients seen in consultation from 12/1/2024-6/1/2025
* Patients aged 18 years to 100 years old
* Patients with a malignancy of breast or head and neck
* English speaking patients
* Patients being treated with definitive intent
* Patients treated at NYU Langone Health for their malignancy
* Willing and able to provide consent

Caregivers:

* Any adult caregiver(s) (aged 18 years to 100 years old) to a patient who fulfills the inclusion and exclusion criteria above.
* Willing and able to provide consent

Providers:

* Doctors and nurse practitioners in medical oncology and radiation oncology, and in the ear nose throat (ENT) department.
* Willing and able to provide consent
* aged 18 years to 100 years old

Exclusion Criteria:

Patients:

* Patients with any other site of disease other than listed above
* Non-English-speaking patients, as the tool is currently available in English only. Translation into additional languages such as Spanish and Russian is currently in process.
* Patient unable to complete the survey portion of the study independently

Caregivers:

• Unable to complete the survey portion of the study independently

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-04-14 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of "Satisfied" Patients | Day 0
  Patients will take a 9-item survey assessing satisfaction with the intervention. Each item is rated as "Yes" or "No." The total score is the sum of "Yes" responses; patients with 6 or more "Yes" answers out of 9 questions are defined as "Satisfied" patients.

SECONDARY OUTCOMES:
Percentage of "Satisfied" Caregivers | Day 0
  Caregivers of patients (if applicable) will take a 10-item survey assessing satisfaction with the intervention. Each item is rated as "Yes" or "No." The total score is the sum of "Yes" responses; caregivers with 7 or more "Yes" answers out of 10 questions will be defined as "Satisfied" caregivers.
Percentage of "Satisfied" Providers | Day 0
  For each patient encountered, providers will take a 5-item survey assessing satisfaction with the intervention. Each item is rated as "Yes" or "No." The total score is the sum of "Yes" responses; a provider with 3 or more "Yes" answers out of 5 questions for a patient will be defined as a "Satisfied" provider for this patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Domogauer, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Jason.Domogauer@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Jason.Domogauer@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.